CLINICAL TRIAL: NCT04645966
Title: A PHASE 2b TRIAL TO ASSESS THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF MenABCWY IN HEALTHY INFANTS 2 AND 6 MONTHS OF AGE
Brief Title: A Clinical Trial to Assess the Safety, Tolerability and Immunogenicity of MenABCWY in Healthy Infants
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Sponsor decided to discontinue the study based on Sponsor's careful review of available safety data in concert with the recommendation of an independent Data Monitoring Committee.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: C3511002; 2020-000948-60 (EudraCT Number)
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Results first posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2023-09

CONDITIONS: Meningococcal Vaccine
Keywords: Meningococcal Vaccine; Invasive Meningococcal Disease; Meningococcal Serogroups A, B, C W and Y; MenABCWY Vaccine
MeSH Terms: interventions — 4CMenB vaccine

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: Open label for Groups 1-5,7,8,10 and 11, no masking; Groups 13-14 is blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- MenABCWY with PLP - 6 months of age (Experimental): Group 1 - Participants 6 months of age vaccinated with MenABCWY on a 2+1 (2 primary vaccinations and a booster dose) schedule, and given Prophylactic Liquid Paracetamol (PLP) during primary vaccinations.
  Interventions: Biological: MenABCWY; Drug: Prophylactic Liquid Paracetamol (PLP)
- MenABCWY - 6 months of age (Experimental): Group 2 - Participants 6 months of age vaccinated with MenABCWY on a 2+1 schedule
  Interventions: Biological: MenABCWY
- Bivalent rLP2086 (60-µg Dose) and Nimerix, with PLP or SLP - 2 months of age (Experimental): Group 3 - Participants 2 months of age vaccinated with Bivalent rLP2086 (60-µg Dose) and Nimenrix on a 2+1 schedule, with PLP or Scheduled Liquid Pracetamol (SLP) during primary vaccinations.
  Interventions: Biological: Bivalent rLP2086 (60-µg Dose); Drug: Prophylactic Liquid Paracetamol (PLP); Biological: Nimenrix; Drug: Scheduled Liquid Paracetamol (SLP)
- Bivalent rLP2086 (60-µg Dose) and Nimenrix - 2 months of age (Experimental): Group 4 - Participants 2 months of age vaccinated with Bivalent rLP2086 (60-mcg Dose) and Nimenrix on a 2+1 schedule
  Interventions: Biological: Bivalent rLP2086 (60-µg Dose); Biological: Nimenrix
- Bivalent rLP2086 (120-µg Dose) and Nimenrix, with PLP - 2 months of age (Experimental): Group 5 - Participants 2 months of age vaccinated with Bivalent rLP2086 (120-µg Dose) and Nimenrix on a 2+1 schedule, and given PLP during primary vaccinations.
  Interventions: Biological: Bivalent rLP2086 (120-µg Dose); Drug: Prophylactic Liquid Paracetamol (PLP); Biological: Nimenrix
- MenABCWY with SLP - 2 months of age (Experimental): Group 7 - Participants 2 months of age vaccinated with MenABCWY on a 2+1 schedule, and given SLP during primary vaccinations.
  Interventions: Biological: MenABCWY; Drug: Scheduled Liquid Paracetamol (SLP)
- Bexsero and Nimenrix with PLP - 2 months of age (Experimental): Group 8 - Participants 2 months of age vaccinated with Bexsero and Nimenrix on a 2+1 schedule, and given PLP during primary vaccinations
  Interventions: Biological: Bexsero; Drug: Prophylactic Liquid Paracetamol (PLP); Biological: Nimenrix
- Bexsero and Nimenrix - 2 months of age (Experimental): Group 10 - Participants 2 months of age vaccinated with Bexsero and Nimenrix on a 2+1 schedule
  Interventions: Biological: Bexsero; Biological: Nimenrix
- MenABCWY with TLP - 2 months of age (Experimental): Group 11 - Participants 2 months of age vaccinated with MenABCWY on a 2+1 schedule, with Therapeutic Liquid Paracetamol (TLP) during primary vaccinations.
  Interventions: Biological: MenABCWY; Drug: Therapeutic Liquid Paracetamol (TLP)
- Blinded: MenABCWY and placebo with SLP or TLP - 2 months of age (Experimental): Group 13 - Participants 2 months of age vaccinated with MenABCWY and placebo on a 2+1 schedule, with a determined ratio of participants given SLP or TLP during primary vaccinations.
  Interventions: Biological: MenABCWY; Other: Placebo; Drug: Scheduled Liquid Paracetamol (SLP); Drug: Therapeutic Liquid Paracetamol (TLP)
- Blinded: Bexsero and Nimenrix with PLP or TLP - 2 months of age (Experimental): Group 14 - Participants 2 months of age vaccinated with Bexsero and Nimenrix on a 2+1 schedule with a determined ratio of participants given PLP or TLP during primary vaccinations.
  Interventions: Biological: Bexsero; Drug: Prophylactic Liquid Paracetamol (PLP); Biological: Nimenrix; Drug: Therapeutic Liquid Paracetamol (TLP)

INTERVENTIONS:
Biological: MenABCWY — Neisseria meningitis groups A, B, C W, and Y vaccine
  Arms: Blinded: MenABCWY and placebo with SLP or TLP - 2 months of age; MenABCWY - 6 months of age; MenABCWY with PLP - 6 months of age; MenABCWY with SLP - 2 months of age; MenABCWY with TLP - 2 months of age
Biological: Bivalent rLP2086 (60-µg Dose) — Trumenba (half dose) - Meningococcal Group B vaccine
  Arms: Bivalent rLP2086 (60-µg Dose) and Nimenrix - 2 months of age; Bivalent rLP2086 (60-µg Dose) and Nimerix, with PLP or SLP - 2 months of age
Biological: Bivalent rLP2086 (120-µg Dose) — Trumenba - Meningococcal Group B vaccine
  Arms: Bivalent rLP2086 (120-µg Dose) and Nimenrix, with PLP - 2 months of age
Biological: Bexsero — Bexsero - Meningococcal Group B vaccine
  Arms: Bexsero and Nimenrix - 2 months of age; Bexsero and Nimenrix with PLP - 2 months of age; Blinded: Bexsero and Nimenrix with PLP or TLP - 2 months of age
Drug: Prophylactic Liquid Paracetamol (PLP) — PLP administration during primary vaccinations 1 and 2
  Arms: Bexsero and Nimenrix with PLP - 2 months of age; Bivalent rLP2086 (120-µg Dose) and Nimenrix, with PLP - 2 months of age; Bivalent rLP2086 (60-µg Dose) and Nimerix, with PLP or SLP - 2 months of age; Blinded: Bexsero and Nimenrix with PLP or TLP - 2 months of age; MenABCWY with PLP - 6 months of age
Biological: Nimenrix — Nimenrix - Meningococcal Group A, C, W and Y vaccine
  Arms: Bexsero and Nimenrix - 2 months of age; Bexsero and Nimenrix with PLP - 2 months of age; Bivalent rLP2086 (120-µg Dose) and Nimenrix, with PLP - 2 months of age; Bivalent rLP2086 (60-µg Dose) and Nimenrix - 2 months of age; Bivalent rLP2086 (60-µg Dose) and Nimerix, with PLP or SLP - 2 months of age; Blinded: Bexsero and Nimenrix with PLP or TLP - 2 months of age
Other: Placebo — Normal Saline
  Arms: Blinded: MenABCWY and placebo with SLP or TLP - 2 months of age
Drug: Scheduled Liquid Paracetamol (SLP) — SLP administration after primary vaccinations 1 and 2.
  Arms: Bivalent rLP2086 (60-µg Dose) and Nimerix, with PLP or SLP - 2 months of age; Blinded: MenABCWY and placebo with SLP or TLP - 2 months of age; MenABCWY with SLP - 2 months of age
Drug: Therapeutic Liquid Paracetamol (TLP) — TLP administration after primary vaccinations 1 and 2
  Arms: Blinded: Bexsero and Nimenrix with PLP or TLP - 2 months of age; Blinded: MenABCWY and placebo with SLP or TLP - 2 months of age; MenABCWY with TLP - 2 months of age

SUMMARY:
The aim of the study is to describe the safety, tolerability, and immunogenicity of MenABCWY in healthy infants 2 and 6 months of age.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants, 2 months of age (≥60 to ≤98 days) or 6 months of age (≥150 to ≤210 days) at the time of randomization.
2. Participant's parent(s)/legal guardian who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.
3. Participant is available for the entire study period and the participant's parent(s)/legal guardian can be reached by telephone.
4. Healthy participant as determined by medical history, physical examination, and judgment of the investigator.
5. Body weight ≥4 kg for participants 2 months of age at the time of randomization.
6. Participants whose parent(s)/legal guardian are capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria:

1. Prior adverse reaction to paracetamol use, including allergic reactions.
2. Participant was born prematurely (<37 weeks of gestation).
3. A previous anaphylactic reaction to any vaccine or vaccine-related component.
4. Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection.
5. A known or suspected defect of the immune system that would prevent an immune response to the vaccine, such as participants with congenital or acquired defects in B-cell function, those receiving chronic systemic (oral, intravenous, or intramuscular) corticosteroid therapy, or those receiving immunosuppressive therapy. Please refer to the SRM for additional details.
6. History of microbiologically proven disease caused by N meningitidis or Neisseria gonorrhoeae.
7. Significant neurological disorder or history of seizure (including simple febrile seizure).
8. Any neuroinflammatory or autoimmune condition, including, but not limited to, transverse myelitis, uveitis, optic neuritis, and multiple sclerosis.
9. Other acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
10. Previous vaccination with any meningococcal vaccine. Written vaccination history must be obtained prior to randomization.
11. For participants 2 months of age, prior vaccination with any of the following licensed or investigational vaccines: pneumococcal vaccine and hexavalent DTPa-HBV-IPV-Hib or its component, except for the birth dose of hepatitis B vaccine.
12. Participants receiving any allergen immunotherapy with a nonlicensed product or receiving allergen immunotherapy with a licensed product and are not on stable maintenance doses.
13. Receipt of any blood products, including immunoglobulin, before the first study vaccination.
14. Current chronic use of systemic antibiotics.
15. Participation in other studies involving investigational drug(s) or investigational vaccine(s) within 28 days prior to study entry and/or during study participation.

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 326 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (21):
- Dr. med Falko Panzer Praxis fuer Kinder und Jugendliche, Mannheim, Germany
- Greece (3):
  - P. & A. Kyriakou Children's Hospital, Athens
  - University General Hospital "ATTIKON", Athens
  - "Ippokratio" General Hospital of Thessaloniki, Thessaloniki
- Spain (17):
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela, A Coruna
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario de Burgos, Burgos, Castille and León
  - Hospital Universitario HM Puerta del Sur, Móstoles, Madrid
  - Centro de Salud L'Eliana, L'Eliana, Valencia
  - Centro de Salud de Paiporta, Paiporta, Valencia
  - Hospital Vithas Virgen del Mar, Almería
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Grupo Pediatrico Uncibay, Málaga
  - Instituto Hispalense de Pediatria, Seville
  - Hospital Universitario Virgen Del Rocio, Seville
  - FISABIO, Valencia
  - Centro de Salud la Serreria II, Valencia
  - Centro de Salud Nazaret, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3511002

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 326 participants signed the informed consent form and were enrolled in the study. Out of which 1 participant was not vaccinated as parent withdrew consent. 325 participants received vaccination. The Sponsor decided to discontinue the study based on Sponsor's careful review of available safety data in concert with the recommendation of an independent Data Monitoring Committee.
Groups:
- Group 1 (MenABCWY +PLP): Infant participants aged 6 months were administered a single intramuscular injection of 0.5 milliliter (mL) Neisseria meningitidis group A, B, C, W, and Y vaccine (MenABCWY) into left thigh at Day 1 (primary vaccination 1) and Month 2 (primary vaccination 2). Prophylactic liquid paracetamol regimen (PLP) was administered orally with 3 required doses, the first dose starting 30 minutes before vaccination (Day 1 [primary vaccination {vacc}1] and Month 2 [primary vaccination 2]). Participants received a single intramuscular injection of MenABCWY approximately 6 months after vaccination 1 (booster vaccination). All participants received a single intramuscular injection of Prevenar 13 and Vaxelis into right thigh on Day 1.
- Group 2 (MenABCWY): Infant participants aged 6 months were administered a single intramuscular injection of 0.5 mL MenABCWY into the left thigh at Day 1 (primary vaccination 1) and Month 2 (primary vaccination 2). Participants received a single intramuscular injection of MenABCWY approximately 6 months after vaccination 1 (booster vaccination). All subjects received a single intramuscular injection of Prevenar 13 and Vaxelis into the right thigh at Day 1.
- Group 3 (60 mcg rLP2086 +Nimenrix +PLP/SLP): Infant participants aged 2 months were administered a single intramuscular injection of 0.25 mL bivalent rLP2086 (60 microgram [mcg]) into the left thigh and 0.5 mL of Nimenrix into the right thigh at Day 1 (primary vaccination 1) and Month 2 (primary vaccination 2). PLP or SLP was administered orally. Participants received a single intramuscular injection of 0.25 mL bivalent rLP2086 (60 mcg) into the left thigh and 0.5 mL of Nimenrix into the right thigh approximately 10 months after vaccination 1 (booster vaccination). All participants received a single intramuscular injection of Prevenar 13 and Vaxelis into the right thigh at 2 and 4 months of age.
- Group 4 (60 mcg rLP2086 +Nimenrix): Infant participants aged 2 months were administered a single intramuscular injection of 0.25 mL of bivalent rLP2086 (60 mcg) into the left thigh and 0.5 mL of Nimenrix into the right thigh at Day 1 (primary vaccination 1) and Month 2 (primary vaccination 2). Participants received a single intramuscular injection of 0.25 mL of bivalent rLP2086 (60 mcg) into the left thigh and 0.5 mL of Nimenrix into the right thigh approximately 10 months after vaccination 1 (booster vaccination). All participants received a single intramuscular injection of Prevenar 13 and Vaxelis into the right thigh at 2 and 4 months of age.
- Group 5 (120 mcg rLP2086 +Nimenrix +PLP): Infant participants aged 2 months were administered a single intramuscular injection of 0.5 mL of bivalent rLP2086 (120 mcg) into the left thigh and 0.5 mL of Nimenrix into the right thigh at Day 1 (primary vaccination 1) and Month 2 (primary vaccination 2). PLP was administered orally with 3 required doses, the first dose starting 30 minutes before vaccination at Day 1 and Month 2. Participants received a single intramuscular injection of 0.5 mL of bivalent rLP2086 (120 mcg) into the left thigh and 0.5 mL of Nimenrix into the right thigh approximately 10 months after vaccination 1 (booster vaccination). All participants received a single intramuscular injection of Prevenar 13 and Vaxelis into the right thigh at 2 and 4 months of age.
- Group 7 (MenABCWY +SLP): Infant participants aged 2 months were administered a single intramuscular injection of 0.5 mL MenABCWY into the left thigh. Scheduled liquid paracetamol (SLP) was administered orally at Day 1 (primary vaccination 1) and Month 2 (primary vaccination 2). Participants received a single intramuscular injection of 0.5 mL MenABCWY approximately 10 months after vaccination 1 (booster vaccination). All participants received a single intramuscular injection of Prevenar 13 and Vaxelis into the right thigh at 2 and 4 months of age. No participants received booster dose due to study termination.
- Group 8 (Bexsero +Nimenrix +PLP): Infant participants aged 2 months were administered a single intramuscular injection of 0.5 mL of Bexsero into the left thigh and 0.5 mL of Nimenrix into the right thigh at Day 1 (primary vaccination 1) and Month 2 (primary vaccination 2). PLP was administered orally with 3 required doses, the first dose starting 30 minutes before vaccination at Day 1 and Month 2. Participants received a single intramuscular injection of 0.5 mL of Bexsero into the left thigh and 0.5 mL of Nimenrix into the right thigh approximately 10 months after vaccination 1 (booster vaccination). All participants received a single intramuscular injection of Prevenar 13 and Vaxelis into the right thigh at 2 and 4 months of age.
- Group 10 (Bexsero +Nimenrix): Infant participants aged 2 months were administered a single intramuscular injection of 0.5 mL of Bexsero into the left thigh and 0.5 mL of Nimenrix into the right thigh at Day 1 (primary vaccination 1), Month 2 (primary vaccination 2) and at approximately 10 months after vaccination 1 (booster vaccination). All participants received a single intramuscular injection of Prevenar 13 and Vaxelis into the right thigh at 2 and 4 months of age.
- Group 11 (MenABCWY +TLP): Infant participants aged 2 months were administered a single intramuscular injection of 0.5 mL MenABCWY into the left thigh at Day 1 (primary vaccination 1). Therapeutic Liquid Paracetamol regimen (TLP) was administered orally. No participants received Vaccination 2 and booster dose due to study termination. All participants received a single intramuscular injection of Prevenar 13 and Vaxelis into the right thigh at 2 months of age.
Period: Vaccination Phase
Arm/Group | Group 1 (MenABCWY +PLP) | Group 2 (MenABCWY) | Group 3 (60 mcg rLP2086 +Nimenrix +PLP/SLP) | Group 4 (60 mcg rLP2086 +Nimenrix) | Group 5 (120 mcg rLP2086 +Nimenrix +PLP) | Group 7 (MenABCWY +SLP) | Group 8 (Bexsero +Nimenrix +PLP) | Group 10 (Bexsero +Nimenrix) | Group 11 (MenABCWY +TLP)
Started | 23 | 25 | 36 | 16 | 53 | 50 | 55 | 55 | 12
Primary Vaccination 1 | 23 | 25 | 39 | 16 | 50 | 50 | 55 | 55 | 12
Primary Vaccination 2 | 22 | 25 | 23 | 16 | 50 | 42 | 54 | 55 | 0
Booster Vaccination | 22 | 25 | 22 | 4 | 9 | 0 | 47 | 45 | 0
Completed | 22 | 25 | 20 | 0 | 2 | 0 | 25 | 22 | 0
Not Completed | 1 | 0 | 16 | 16 | 51 | 50 | 30 | 33 | 12
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 14 | 15 | 47 | 43 | 29 | 29 | 12
Not completed — Withdrawal by parent/guardian | 0 | 0 | 2 | 1 | 3 | 4 | 0 | 2 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — No longer meets eligibility criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Follow-up Phase
Arm/Group | Group 1 (MenABCWY +PLP) | Group 2 (MenABCWY) | Group 3 (60 mcg rLP2086 +Nimenrix +PLP/SLP) | Group 4 (60 mcg rLP2086 +Nimenrix) | Group 5 (120 mcg rLP2086 +Nimenrix +PLP) | Group 7 (MenABCWY +SLP) | Group 8 (Bexsero +Nimenrix +PLP) | Group 10 (Bexsero +Nimenrix) | Group 11 (MenABCWY +TLP)
Started | 22 | 25 | 20 | 0 | 2 | 0 | 25 | 22 | 0
Completed | 22 | 25 | 20 | 0 | 2 | 0 | 25 | 21 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least 1 dose of investigational product and had safety data reported after vaccination.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (MenABCWY +PLP) | Group 2 (MenABCWY) | Group 3 (60 mcg rLP2086 +Nimenrix +PLP/SLP) | Group 4 (60 mcg rLP2086 +Nimenrix) | Group 5 (120 mcg rLP2086 +Nimenrix +PLP) | Group 7 (MenABCWY +SLP) | Group 8 (Bexsero +Nimenrix +PLP) | Group 10 (Bexsero +Nimenrix) | Group 11 (MenABCWY +TLP) | Total
Number analyzed (Participants) | 23 | 25 | 36 | 16 | 53 | 50 | 55 | 55 | 12 | 325
Age, Continuous [Mean (Standard Deviation); unit: Days] | 158.5 (6.87) | 161.6 (14.45) | 71.1 (7.00) | 67.6 (5.81) | 68.9 (6.39) | 68.0 (5.99) | 67.4 (7.89) | 67.5 (7.30) | 69.4 (7.69) | 81.9 (33.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 21 | 7 | 24 | 27 | 32 | 20 | 7 | 160
  Male | 11 | 15 | 15 | 9 | 29 | 23 | 23 | 35 | 5 | 165
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 9 | 21 | 8 | 10 | 25 | 18 | 22 | 6 | 132
  Not Hispanic or Latino | 10 | 16 | 15 | 8 | 43 | 25 | 37 | 33 | 6 | 193
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  White | 20 | 24 | 35 | 16 | 52 | 50 | 55 | 55 | 12 | 319
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Serum Bactericidal Assay Using Human Complement (hSBA) Titer >=LLOQ for Each MenA, MenC, MenW and MenY Test Strains 1 Month After Primary Vaccination 2: Group 7 and 11 Combined Versus Group 8 and 10 Combined
Description: Percentage of participants achieving hSBA titer greater than or equal to (>=) lower limit of quantitation (LLOQ) (i.e.,1:8) for each MenA, MenC, MenW and MenY test strains were reported in this outcome measure. Exact 2-sided confidence interval (CI) using the Clopper and Pearson method was presented. Analysis was performed on Post-primary vaccination 2 (post-PV2) evaluable immunogenicity population (EIP). No serum samples collected after vaccination 2 for participants in Group 11 as participants were not administered PV 2 due to study termination.
Time Frame: 1 month after primary vaccination 2
Population: Post-PV 2 EIP: participants randomized,eligible through Visit(V)4;received vaccine at V1,V3;blood drawn for assay test within required timeframes at V4;had at least 1 valid, determinate MenA,C,W,Y,or B assay result at V4;received no prohibited vaccines/treatment,no protocol deviation through V4.''N''=participants evaluable for outcome measure; ''n''=participants evaluable for specific rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Group 7 and 11 Combined: Group 7: Infant participants aged 2 months were administered a single intramuscular injection of 0.5 mL MenABCWY into the left thigh. Scheduled liquid paracetamol (SLP) was administered orally at Day 1 (primary vaccination 1) and Month 2 (primary vaccination 2). All participants received a single intramuscular injection of Prevenar 13 and Vaxelis into the right thigh at 2 and 4 months of age. Group11: Infant participants aged 2 months were administered a single intramuscular injection of 0.5 mL MenABCWY into the left thigh at Day 1 (primary vaccination 1). TLP regimen was administered orally. No serum samples collected after vaccination 2 for participants in Group 11 as participants were not administered PV 2 due to study termination.
- Group 8 and 10 Combined: Infant participants aged 2 months were administered single IM injection of 0.5mL of Bexsero into left thigh, 0.5mL of Nimenrix into right thigh at Day 1(primary vaccination 1), Month 2 (primary vaccination 2) and approximately 10 months after vaccination 1 (booster vaccination). Participants in Group 8 were administered PLP orally with 3 required doses, first dose starting 30 minutes before vaccination at Day1 and Month 2. All participants received single IM injection of Prevenar 13 and Vaxelis into right thigh at 2 and 4 months of age.
Arm/Group | Group 7 and 11 Combined | Group 8 and 10 Combined
Number analyzed (Participants) | 16 | 92
Percentage of participants
  MenA: number analyzed (Participants) | 16 | 90
  MenA | 100.0 [79.4 to 100.0] | 100.0 [96.0 to 100.0]
  MenC: number analyzed (Participants) | 16 | 91
  MenC | 100.0 [79.4 to 100.0] | 100.0 [96.0 to 100.0]
  MenW: number analyzed (Participants) | 16 | 91
  MenW | 100.0 [79.4 to 100.0] | 100.0 [96.0 to 100.0]
  MenY | 100.0 [79.4 to 100.0] | 100.0 [96.1 to 100.0]

2. Primary Outcome: Percentage of Participants Achieving hSBA Titer >= LLOQ for Each MenACWY MenA, MenC, MenW and MenY Test Strains 1 Month After Booster Vaccination: Group 7 and 11 Combined Versus Group 8 and 10 Combined
Description: Percentage of participants achieving hSBA titer >= LLOQ (1:8) for each MenA, MenC, MenW and MenY test strains were reported in this outcome measure. Exact 2-sided CI using the Clopper and Pearson method was presented. No participants in Group 7 and Group 11 received booster vaccination due to study termination.
Time Frame: 1 month after booster vaccination
Population: Post-booster vaccination EIP: randomized participants eligible through V6;received vaccine at V1, V3, V5;blood drawn for assay testing within required timeframes at V6; had at least 1 valid, determinate MenA, MenC, MenW, MenY, or MenB assay result at V6; received no prohibited vaccines/treatment and had no protocol deviations through V6. Here, ''N''=participants evaluable for the outcome measure and ''n''=participants evaluable for specific rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Group 7 and 11 Combined: Group 7: Infant participants aged 2 months were administered a single intramuscular injection of 0.5 mL MenABCWY into the left thigh. Scheduled liquid paracetamol (SLP) was administered orally at Day 1 (primary vaccination 1) and Month 2 (primary vaccination 2). All participants received a single intramuscular injection of Prevenar 13 and Vaxelis into the right thigh at 2 and 4 months of age. Group11: Infant participants aged 2 months were administered a single intramuscular injection of 0.5 mL MenABCWY into the left thigh at Day 1 (primary vaccination 1). TLP regimen was administered orally.
Arm/Group | Group 7 and 11 Combined | Group 8 and 10 Combined
Number analyzed (Participants) | 0 | 42
Percentage of participants
  MenA: number analyzed (Participants) | 0 | 41
  MenA |  | 100.0 [91.4 to 100.0]
  MenC: number analyzed (Participants) | 0 | 41
  MenC |  | 100.0 [91.4 to 100.0]
  MenW |  | 100.0 [91.6 to 100.0]
  MenY: number analyzed (Participants) | 0 | 41
  MenY |  | 100.0 [91.4 to 100.0]

3. Primary Outcome: Percentage of Participants Achieving hSBA Titer >= LLOQ for Each Neisseria Meningitidis Group B (MenB) Test Strain 1 Month After Primary Vaccination 2: Group 7 and 11 Combined Versus Group 8 and 10 Combined
Description: Percentage of participants achieving hSBA titer>= LLOQ for each MenB test strain (1:16 for strain A22 and 1:8 for strain B44) is reported in this outcome measure. Exact 2-sided CI using Clopper and Pearson method is presented. No serum samples collected after vaccination 2 for participants in Group 11 as participants were not administered PV 2 due to study termination.
Time Frame: 1 month After primary vaccination 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 7 and 11 Combined | Group 8 and 10 Combined
Number analyzed (Participants) | 18 | 95
Percentage of participants
  PMB80 (A22): number analyzed (Participants) | 18 | 94
  PMB80 (A22) | 44.4 [21.5 to 69.2] | 9.6 [4.5 to 17.4]
  PMB2707 (B44) | 88.9 [65.3 to 98.6] | 29.5 [20.6 to 39.7]

4. Primary Outcome: Percentage of Participants Achieving hSBA Titer >= LLOQ for Each Neisseria Meningitidis Group B (MenB) Test Strain 1 Month After Primary Vaccination 2: Group 3 and 4 Combined Versus Group 5
Description: Percentage of participants achieving hSBA titer>= LLOQ for each MenB test strain(1:16 for strain A22 and 1:8 for strain B44) is reported in this outcome measure. Exact 2-sided CI using Clopper and Pearson method is presented.
Time Frame: 1 month after primary vaccination 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Group 3 and 4 Combined: Infant participants aged 2 months were administered single IM injection of 0.25mL bivalent rLP2086(60μg) into left thigh,0.5mL Nimenrix into right thigh at Day 1(primary vacc 1),Month 2(primary vacc 2).PLP or SLP administered orally. Participants received single IM injection of 0.25mL bivalent rLP2086(60 μg) into left thigh and 0.5mL Nimenrix into right thigh approx. 10 months after vacc1(booster vacc).Participants received single IM injection of Prevenar 13,Vaxelis into right thigh at 2 and 4 months of age.
Arm/Group | Group 3 and 4 Combined | Group 5 (120 mcg rLP2086 +Nimenrix +PLP)
Number analyzed (Participants) | 35 | 45
Percentage of participants
  PMB80 (A22): number analyzed (Participants) | 30 | 44
  PMB80 (A22) | 46.7 [28.3 to 65.7] | 47.7 [32.5 to 63.3]
  PMB2707 (B44) | 82.9 [66.4 to 93.4] | 97.8 [88.2 to 99.9]

5. Primary Outcome: Percentage of Participants Achieving hSBA Titer >= LLOQ for Each MenB Test Strain 1 Month After Booster Vaccination: Group 7 and 11 Combined Versus Group 8 and 10 Combined
Description: Percentage of participants achieving hSBA titer>= LLOQ for each MenB test strain (1:16 for strain A22 and 1:8 for strain B44) is reported in this outcome measure. Exact 2-sided CI using Clopper and Pearson method is presented. No participants in Group 7 and Group 11 received booster vaccination due to study termination.
Time Frame: 1 Month after booster vaccination
Population: Post booster vacc. evaluable immunogenicity population=randomised to study group of interest,eligible through V6. Received investigational products at V1,3,5 as randomised,blood drawn for assay testing at required time frames at V6(1 month after booster vacc[28-42 days]).At least 1 valid,determinate MenA, C, W, Y,or B assay result at V6, received no prohibited vaccines/treatment, no protocol deviations through V6.''N''=participants evaluable here; ''n''=participants evaluable for specific rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 7 and 11 Combined | Group 8 and 10 Combined
Number analyzed (Participants) | 0 | 41
Percentage of participants
  PMB80 (A22): number analyzed (Participants) | 0 | 40
  PMB80 (A22) |  | 25.0 [12.7 to 41.2]
  PMB2707 (B44) |  | 34.1 [20.1 to 50.6]

6. Primary Outcome: Percentage of Participants Achieving hSBA Titer >= LLOQ for Each MenB Test Strain 1 Month After Booster Vaccination: Groups 3, 4 and 5
Description: Percentage of participants achieving hSBA titer >= LLOQ for each MenB test strain (1:16 for strain A22 and 1:8 for strain B44) is reported in this outcome measure. Exact 2-sided CI using Clopper and Pearson method is presented. Groups 4 and 5 had no serum samples collected post-booster for serology testing due to study termination.
Time Frame: 1 Month after booster vaccination
Population: Post booster vacc. evaluable immunogenicity population=randomised to study group of interest,eligible through V6. Received investigational products at V1,3,5 as randomised,blood drawn for assay testing at required time frames at V6(1 month after booster vacc[28-42 days]).At least 1 valid,determinate MenA, C, W, Y,or B assay result at V6, received no prohibited vaccines/treatment, no protocol deviations through V6.''N''=participants evaluable here.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 3 (60 mcg rLP2086 +Nimenrix +PLP/SLP) | Group 4 (60 mcg rLP2086 +Nimenrix) | Group 5 (120 mcg rLP2086 +Nimenrix +PLP)
Number analyzed (Participants) | 18 | 0 | 0
Percentage of participants
  PMB80 (A22) | 38.9 [17.3 to 64.3] |  |
  PMB2707 (B44) | 83.3 [58.6 to 96.4] |  |

7. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Primary Vaccination 1: Group 7 and 11 Combined Versus Group 8 and 10 Combined
Description: Local reactions included tenderness at injection site, redness and swelling and were recorded by participant's parents/legal guardians in an electronic diary (e-diary). Redness and swelling were measured and recorded in caliper units. 1 caliper unit =0.5 centimeter (cm) and graded as mild: 0.5 to 2.0 cm, moderate: >2.0 to 7.0 cm and severe: >7.0 cm. Tenderness at injection site was graded as mild: hurt if gently touched, moderate: hurt if gently touched with crying and severe: caused limitation of limb movement. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Within 7 days after primary vaccination 1
Population: Primary vaccination 1 safety population included all randomised participants who received the first dose of investigational product at Visit 1 and had safety follow-up between Visit 1 and prior to Visit 3. Here, ''N''=participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 7 and 11 Combined | Group 8 and 10 Combined
Number analyzed (Participants) | 62 | 108
Percentage of participants
  Redness: Mild | 22.6 [12.9 to 35.0] | 23.1 [15.6 to 32.2]
  Redness: Moderate | 11.3 [4.7 to 21.9] | 6.5 [2.6 to 12.9]
  Redness: Severe | 0 [0.0 to 5.8] | 0 [0.0 to 3.4]
  Swelling: Mild | 21.0 [11.7 to 33.2] | 22.2 [14.8 to 31.2]
  Swelling: Moderate | 17.7 [9.2 to 29.5] | 12.0 [6.6 to 19.7]
  Swelling: Severe | 0 [0.0 to 5.8] | 0 [0.0 to 3.4]
  Tenderness at injection site: Mild | 22.6 [12.9 to 35.0] | 25.9 [18.0 to 35.2]
  Tenderness at injection site: Moderate | 48.4 [35.5 to 61.4] | 24.1 [16.4 to 33.3]
  Tenderness at injection site: Severe | 0 [0.0 to 5.8] | 0.9 [0.0 to 5.1]

8. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Primary Vaccination 2: Group 7 Versus Group 8 and 10 Combined
Description: Local reactions included tenderness at injection site, redness and swelling and were recorded by participant's parents/legal guardians in an e-diary. Redness and swelling were measured and recorded in caliper units. 1 caliper unit =0.5 cm and graded as mild: 0.5 to 2.0 cm, moderate: >2.0 to 7.0 cm and severe: >7.0 cm. Tenderness at injection site was graded as mild: hurt if gently touched, moderate: hurt if gently touched with crying and severe: caused limitation of limb movement. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Within 7 Days after primary Vaccination 2
Population: Primary vaccination 2 safety population included all participants who received the second dose of investigational product at Visit 3 and who had safety follow-up between Visit 3 and prior to Visit 4. Here, ''N''=participants evaluable for this outcome measure. Data was not collected from participants in Group 11 as no participants received primary vaccination 2 due to study termination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Group 7: Group 7: Infant participants aged 2 months were administered a single intramuscular injection of 0.5 mL MenABCWY into the left thigh. Scheduled liquid paracetamol (SLP) was administered orally at Day 1 (primary vaccination 1) and Month 2 (primary vaccination 2). All participants received a single intramuscular injection of Prevenar 13 and Vaxelis into the right thigh at 2 and 4 months of age.
- Group 8 and 10 Combined: Group8:Infant participants aged 2 months were administered single IM injection of 0.5mL of Bexsero into left thigh, 0.5mL of Nimenrix into right thigh at Day 1(primary vaccination 1) and Month 2(primary vaccination 2).PLP was administered orally with 3 required doses,first dose starting 30 minutes before vaccination at Day1 and Month2.Participants received single IM injection of 0.5mL of Bexsero into left thigh and 0.5mL of Nimenrix into right thigh approximately 10 months after vaccination 1 (booster vaccination).Participants received single IM injection of Prevenar 13 and Vaxelis into right thigh at 2,4 months of age.Group10:Infant participants aged 2 months were administered single IM injection of 0.5mL of Bexsero into left thigh,0.5mL of Nimenrix into right thigh at Day 1(primary vaccination 1), Month 2(primary vaccination 2) and approximately 10 months after vaccination1 (booster vaccination).Participants received single IM injection of Prevenar 13 and Vaxelis into right thigh at 2,4 months of age.
Arm/Group | Group 7 | Group 8 and 10 Combined
Number analyzed (Participants) | 41 | 107
Percentage of participants
  Redness: Mild | 26.8 [14.2 to 42.9] | 27.1 [19.0 to 36.6]
  Redness: Moderate | 12.2 [4.1 to 26.2] | 11.2 [5.9 to 18.8]
  Redness: Severe | 0 [0.0 to 8.6] | 0 [0.0 to 3.4]
  Swelling: Mild | 19.5 [8.8 to 34.9] | 25.2 [17.3 to 34.6]
  Swelling: Moderate | 14.6 [5.6 to 29.2] | 12.1 [6.6 to 19.9]
  Swelling: Severe | 0 [0.0 to 8.6] | 0 [0.0 to 3.4]
  Tenderness at injection site: Mild | 22.0 [10.6 to 37.6] | 27.1 [19.0 to 36.6]
  Tenderness at injection site: Moderate | 34.1 [20.1 to 50.6] | 23.4 [15.7 to 32.5]
  Tenderness at injection site: Severe | 4.9 [0.6 to 16.5] | 2.8 [0.6 to 8.0]

9. Primary Outcome: Percentage of Participants With Systemic Events and Antipyretic Use Within 7 Days After Primary Vaccination 1: Group 7 and 11 Combined Versus Group 8 and 10 Combined
Description: Systemic events were recorded by participant's parents/legal guardians in e-diary. Fever was defined as temperature >=38.0 degrees (deg) Celsius(C) and was categorized as 38.0 to 38.4 deg C, >38.4 to 38.9 deg C, >38.9 to 40.0 deg C and >40.0 deg C. Decreased appetite was categorized as Mild: decreased interest in eating, Moderate: decreased oral intake, Severe: refusal to feed. Drowsiness: Mild: Increased or prolonged sleeping bouts, Moderate: Slightly subdued interfering with daily activity, Severe; Disabling, not interested in usual daily activity. Irritability; Mild: Easily consolable, Moderate: required increased attention, Severe: Inconsolable; crying could not be comforted. Exact 2-sided CI was based on the Clopper and Pearson method
Time Frame: Within 7 Days after primary Vaccination 1
Population: Primary vaccination 1 safety population included all randomized participants who received the first dose of investigational product at Visit 1 and had safety follow-up between Visit 1 and prior to Visit 3. Here, ''N''=participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 7 and 11 Combined | Group 8 and 10 Combined
Number analyzed (Participants) | 62 | 108
Percentage of participants
  Fever: 38.0°C to 38.4°C | 29.0 [18.2 to 41.9] | 15.7 [9.4 to 24.0]
  Fever: >38.4°C to 38.9°C | 24.2 [14.2 to 36.7] | 5.6 [2.1 to 11.7]
  Fever: >38.9°C to 40.0°C | 9.7 [3.6 to 19.9] | 0 [0.0 to 3.4]
  Fever: >40.0°C | 0 [0.0 to 5.8] | 0 [0.0 to 3.4]
  Decreased appetite: Mild | 17.7 [9.2 to 29.5] | 17.6 [10.9 to 26.1]
  Decreased appetite: Moderate | 43.5 [31.0 to 56.7] | 21.3 [14.0 to 30.2]
  Decreased appetite: Severe | 4.8 [1.0 to 13.5] | 0.9 [0.0 to 5.1]
  Irritability: Mild | 21.0 [11.7 to 33.2] | 19.4 [12.5 to 28.2]
  Irritability: Moderate | 59.7 [46.4 to 71.9] | 45.4 [35.8 to 55.2]
  Irritability: Severe | 14.5 [6.9 to 25.8] | 6.5 [2.6 to 12.9]
  Drowsiness: Mild | 37.1 [25.2 to 50.3] | 39.8 [30.5 to 49.7]
  Drowsiness: Moderate | 32.3 [20.9 to 45.3] | 18.5 [11.7 to 27.1]
  Drowsiness: Severe | 4.8 [1.0 to 13.5] | 0.9 [0.00 to 5.1]
  Use of antipyretic medication | 46.8 [34.0 to 59.9] | 50.0 [40.2 to 59.8]

10. Primary Outcome: Percentage of Participants With Systemic Events and Antipyretic Use Within 7 Days After Primary Vaccination 2: Group 7 Versus Group 8 and 10 Combined
Description: Systemic events were recorded by participant's parents/legal guardians in e-diary. Fever was defined as temperature >=38.0 deg C and was categorized as 38.0 to 38.4 deg C, >38.4 to 38.9 deg C, >38.9 to 40.0 deg C and >40.0 deg C. Decreased appetite was categorized as Mild: decreased interest in eating, Moderate: decreased oral intake, Severe: refusal to feed. Drowsiness was graded as Mild: Increased or prolonged sleeping bouts, Moderate: Slightly subdued interfering with daily activity, Severe; Disabling, not interested in usual daily activity. Irritability; Mild: Easily consolable, Moderate: required increased attention, Severe: Inconsolable; crying could not be comforted. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Within 7 days after primary vaccination 2
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Group 7: Group7: Infant participants aged 2 months were administered a single intramuscular injection of 0.5 mL MenABCWY into the left thigh. Scheduled liquid paracetamol (SLP) was administered orally at Day 1 (primary vaccination 1) and Month 2 (primary vaccination 2). Participants received a single intramuscular injection of 0.5 mL MenABCWY approximately 10 months after vaccination 1 (booster vaccination). All participants received a single intramuscular injection of Prevenar 13 and Vaxelis into the right thigh at 2 and 4 months of age.
Arm/Group | Group 7 | Group 8 and 10 Combined
Number analyzed (Participants) | 41 | 107
Percentage of participants
  Fever: 38.0°C to 38.4°C | 26.8 [14.2 to 42.9] | 31.8 [23.1 to 41.5]
  Fever: >38.4°C to 38.9°C | 26.8 [14.2 to 42.9] | 14.0 [8.1 to 22.1]
  Fever: >38.9°C to 40.0°C | 12.2 [4.1 to 26.2] | 2.8 [0.6 to 8.0]
  Fever: >40.0°C | 0 [0.0 to 8.6] | 0 [0.0 to 3.4]
  Decreased appetite: Mild | 22.0 [10.6 to 37.6] | 20.6 [13.4 to 29.5]
  Decreased appetite: Moderate | 31.7 [18.1 to 48.1] | 25.2 [17.3 to 34.6]
  Decreased appetite: Severe | 4.9 [0.6 to 16.5] | 3.7 [1.0 to 9.3]
  Irritability: Mild | 12.2 [4.1 to 26.2] | 21.5 [14.1 to 30.5]
  Irritability: Moderate | 53.7 [37.4 to 69.3] | 48.6 [38.8 to 58.5]
  Irritability: Severe | 22.0 [10.6 to 37.6] | 6.5 [2.7 to 13.0]
  Drowsiness: Mild | 29.3 [16.1 to 45.5] | 45.8 [36.1 to 55.7]
  Drowsiness: Moderate | 34.1 [20.1 to 50.6] | 14.0 [8.1 to 22.1]
  Drowsiness: Severe | 4.9 [0.6 to 16.5] | 0.9 [0.0 to 5.1]
  Use of antipyretic medication | 41.5 [26.3 to 57.9] | 72.9 [63.4 to 81.0]

11. Primary Outcome: Percentage of Participants With AEs, SAEs, MAEs and NDCMC Within 30 Days After Primary Vaccination 1: Group 7 and 11 Combined Versus Group 8 and 10 Combined
Description: An adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of investigational product, whether or not considered related to the investigational product. A serious adverse event (SAE) was any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent disability/incapacity; congenital anomaly/birth defect and other important medical events. Medically attended adverse event (MAE) was defined as a nonserious AE that resulted in an evaluation at a medical facility. Newly diagnosed chronic medical condition (NDCMC) was defined as a disease or medical condition, not previously identified, that was expected to be persistent or otherwise long-lasting in its effects.
Time Frame: Within 30 days after primary vaccination 1
Population: Safety population included all randomized participants who received at least 1 dose of investigational product and had safety data reported after vaccination. Here, ''N''=participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 7 and 11 Combined | Group 8 and 10 Combined
Number analyzed (Participants) | 62 | 110
Percentage of participants
  AEs | 24.2 | 16.4
  SAEs | 4.8 | 0
  MAEs | 14.5 | 10.0
  NDCMCs | 0 | 0.9

12. Primary Outcome: Percentage of Participants With AEs, SAEs,MAEs and NDCMC Within 30 Days After Primary Vaccination 2: Group 7 Versus Group 8 and 10 Combined
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of investigational product, whether or not considered related to the investigational product. An SAE was any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent disability/incapacity; congenital anomaly/birth defect and other important medical events. MAE was defined as a nonserious AE that resulted in an evaluation at a medical facility. NDCMC was defined as a disease or medical condition, not previously identified, that wasis expected to be persistent or otherwise long-lasting in its effects.
Time Frame: Within 30 days after primary vaccination 2
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | Group 7 | Group 8 and 10 Combined
Number analyzed (Participants) | 42 | 109
Percentage of participants
  AEs | 33.3 | 12.8
  SAEs | 2.4 | 0
  MAEs | 23.8 | 11.0
  NDCMC | 0 | 0.9

13. Primary Outcome: Percentage of Participants With AEs, SAEs, MAEs and NDCMC Within 30 Days After Any Primary Vaccination: Group 7 and 11 Combined Versus Group 8 and 10 Combined
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of investigational product, whether or not considered related to the investigational product. An SAE was any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent disability/incapacity; congenital anomaly/birth defect and other important medical events. MAE was defined as a nonserious AE that resulted in an evaluation at a medical facility. NDCMC was defined as a disease or medical condition, not previously identified, that is was expected to be persistent or otherwise long-lasting in its effects.
Time Frame: Within 30 days after any primary vaccination
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Group 7 and 11 Combined | Group 8 and 10 Combined
Number analyzed (Participants) | 62 | 110
Percentage of participants
  AEs | 40.3 | 24.5
  SAEs | 6.5 | 0
  MAEs | 29.0 | 16.4
  NDCMC | 0 | 0.9

14. Primary Outcome: Percentage of Participants With AEs, SAEs, MAEs and NDCMC During Primary Series Vaccination Phase: Group 7 and 11 Combined Versus Group 8 and 10 Combined
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of investigational product, whether or not considered related to the investigational product. SAE was any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent disability/incapacity; congenital anomaly/birth defect and other important medical events. MAE was defined as a nonserious AE that resulted in an evaluation at a medical facility. NDCMC was defined as a disease or medical condition, not previously identified, that was expected to be persistent or otherwise long-lasting in its effects.
Time Frame: From day of primary vaccination 1 at Day 1 up to 1 month after primary vaccination 2
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Group 7 and 11 Combined | Group 8 and 10 Combined
Number analyzed (Participants) | 62 | 110
Percentage of participants
  AEs | 56.5 | 33.6
  SAEs | 6.5 | 1.8
  MAEs | 43.5 | 24.5
  NDCMC | 1.6 | 0.9

15. Primary Outcome: Percentage of Participants With SAEs, MAEs and NDCMC During Primary Series Follow-up Phase: Group 7 Versus Group 8 and 10 Combined
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of investigational product, whether or not considered related to the investigational product. An SAE was any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent disability/incapacity; congenital anomaly/birth defect and other important medical events. MAE was defined as a nonserious AE that resulted in an evaluation at a medical facility. NDCMC was defined as a disease or medical condition, not previously identified, that was expected to be persistent or otherwise long-lasting in its effects.
Time Frame: From 1 month after primary vaccination 2 up to booster vaccination
Population: Safety population included all randomized participants who received at least 1 dose of investigational product and had safety data reported after vaccination. Here, ''N''=participants evaluable for this outcome measure. Data was not collected from participants in Group 11 as no participants received primary vaccination 2 due to study termination.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 7 | Group 8 and 10 Combined
Number analyzed (Participants) | 41 | 109
Percentage of participants
  AEs | 17.1 | 18.3
  SAEs | 4.9 | 2.8
  MAEs | 12.2 | 15.6
  NDCMC | 0 | 0.9

16. Primary Outcome: Percentage of Participants With AEs, SAEs, MAEs and NDCMC Throughout Primary Series Stage: Group 7 and 11 Combined Versus Group 8 and 10 Combined
Description: Infant participants aged 2 months were administered single IM injection of 0.5mL of Bexsero into left thigh, 0.5mL of Nimenrix into right thigh at Day 1(primary vaccination 1), Month 2 (primary vaccination 2) and approximately 10 months after vaccination 1 (booster vaccination). Participants in Group 8 were administered PLP orally with 3 required doses, first dose starting 30 minutes before vaccination at Day1 and Month 2. All participants received single IM injection of Prevenar 13 and Vaxelis into right thigh at 2 and 4 months of age.
Time Frame: From the date of primary vaccination 1 up to 8 months after primary vaccination 2 (maximum up to 9 months)
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Group 7 and 11 Combined | Group 8 and 10 Combined
Number analyzed (Participants) | 62 | 110
Percentage of participants
  AEs | 59.7 | 40.0
  SAEs | 9.7 | 4.5
  MAEs | 45.2 | 30.0
  NDCMC | 1.6 | 1.8

17. Primary Outcome: Percentage of Participants With Immediate AEs Within 30 Minutes After Primary Vaccination 1: Groups 7 and 11 Combined Versus Groups 8 and 10 Combined
Description: Immediate AEs were defined as AEs occurring within the first 30 minutes after investigational product administration.
Time Frame: Within 30 minutes After primary vaccination 1
Population: Primary vaccination 1 safety population included all participants who received the first dose of investigational product at Visit 1 and who had safety follow-up between Visit 1 and prior to Visit 3. Here, ''N''=participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 7 and 11 Combined | Group 8 and 10 Combined
Number analyzed (Participants) | 62 | 110
Percentage of participants | 0 | 0

18. Primary Outcome: Percentage of Participants With Immediate AEs Within 30 Minutes After Primary Vaccination 2: Group 7 Versus Groups 8 and 10 Combined
Description: Immediate AEs were defined as AEs occurring within the first 30 minutes after investigational product administration.
Time Frame: Within 30 minutes After primary vaccination 2
Population: Primary vaccination 2 safety population included all participants who received the second dose of investigational product at Visit 3 and who had safety follow-up between Visit 3 and prior to Visit 4. Here, ''N''=participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 7 | Group 8 and 10 Combined
Number analyzed (Participants) | 42 | 109
Percentage of participants | 0 | 0

19. Primary Outcome: Percentage of Participants With Immediate AEs After Booster Vaccination: Group 7 and 11 Combined Versus Group 8 and 10 Combined
Description: Immediate AEs were defined as AEs occurring within the first 30 minutes after investigational product administration.
Time Frame: Within 30 minutes after booster vaccination
Population: Booster vaccination safety population included participants who received booster dose of investigational product, had safety follow-up between Visit 5 and prior to Visit 6 (after booster vaccination). Here, 'N'=participants evaluable for this outcome measure. Data was not collected from participants in Groups 7 and 11 as no participants received booster vaccination due to study termination.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 7 and 11 Combined | Group 8 and 10 Combined
Number analyzed (Participants) | 0 | 92
Percentage of participants |  | 0

20. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Booster Vaccination: Group 7 and 11 Combined Versus Group 8 and 10 Combined
Description: Local reactions included tenderness at injection site, redness and swelling and were recorded by participant's parents/legal guardians in an electronic diary (e-diary). Redness and swelling were measured and recorded in caliper units. 1 caliper unit =0.5 centimeter (cm) and graded as mild: 0.5 to 2.0 cm, moderate: >2.0 to 7.0 cm and severe: >7.0 cm. Tenderness at injection site was graded as mild: hurt if gently touched, moderate: hurt if gently touched with crying and severe: caused limitation of limb movement.
Time Frame: Within 7 Days after booster vaccination
Population: as for outcome 19
Measure: Number; unit: Participants
Arm/Group | Group 7 and 11 Combined | Group 8 and 10 Combined
Number analyzed (Participants) | 0 | 92
Participants
  Redness |  | 38
  Swelling |  | 35
  Tenderness at injection site |  | 63

21. Primary Outcome: Percentage of Participants With Systemic Events and Antipyretic Use Within 7 Days After Booster Vaccination: Group 7 and 11 Combined Versus Group 8 and 10 Combined
Description: Systemic events were recorded by participant's parents/legal guardians in e-diary. Fever was defined as temperature >=38.0 deg C, categorized as 38.0 to 38.4 deg C, >38.4 to 38.9 deg C, >38.9 to 40.0 deg C and >40.0 deg C. Decreased appetite was graded as Mild: decreased interest in eating, Moderate: decreased oral intake, Severe: refusal to feed. Drowsiness: Mild: Increased or prolonged sleeping bouts, Moderate: Slightly subdued interfering with daily activity, Severe; Disabling, not interested in usual daily activity. Irritability; Mild: Easily consolable, Moderate: required increased attention, Severe: Inconsolable; crying could not be comforted. Exact 2-sided CI was based on Clopper and Pearson method.
Time Frame: Within 7 days after booster vaccination
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 7 and 11 Combined | Group 8 and 10 Combined
Number analyzed (Participants) | 0 | 91
Percentage of participants
  Fever: 38.0°C to 38.4°C |  | 19.8 [12.2 to 29.4]
  Fever: >38.4°C to 38.9°C |  | 11.0 [5.4 to 19.3]
  Fever: >38.9°C to 40.0°C |  | 4.4 [1.2 to 10.9]
  Fever: >40.0°C |  | 0 [0.0 to 4.0]
  Decreased appetite: Mild |  | 17.6 [10.4 to 27.0]
  Decreased appetite: Moderate |  | 27.5 [18.6 to 37.8]
  Decreased appetite: Severe |  | 2.2 [0.3 to 7.7]
  Irritability: Mild |  | 22.0 [14.0 to 31.9]
  Irritability: Moderate |  | 42.9 [32.5 to 53.7]
  Irritability: Severe |  | 7.7 [3.1 to 15.2]
  Drowsiness: Mild |  | 26.4 [17.7 to 36.7]
  Drowsiness: Moderate |  | 18.7 [11.3 to 28.2]
  Drowsiness: Severe |  | 1.1 [0.0 to 6.0]
  Use of antipyretic medication |  | 63.7 [53.0 to 73.6]

22. Primary Outcome: Percentage of Participants With AEs, SAEs, MAEs and NDCMC During Booster Vaccination Phase: Group 7 and 11 Combined Versus Group 8 and 10 Combined
Description: as for outcome 15
Time Frame: From date of booster vaccination through 1 month after booster vaccination
Population: as for outcome 19
Measure: Number; unit: Percentage of participants
Arm/Group | Group 7 and 11 Combined | Group 8 and 10 Combined
Number analyzed (Participants) | 0 | 92
Percentage of participants
  AEs |  | 27.2
  SAEs |  | 0
  MAEs |  | 92
  NDCMC |  | 0

23. Primary Outcome: Percentage of Participants With AEs, SAEs, MAEs and NDCMC During Booster Follow-up Phase: Group 7 and 11 Combined Versus Group 8 and 10 Combined
Description: as for outcome 15
Time Frame: From 1 month after booster vaccination up to 6 months after booster vaccination (maximum up to 5 months)
Population: Booster vaccination follow-up safety population included participants who received the booster dose of investigational product and who had safety follow-up between Visit 6 and up to and including Visit 7 (after booster vaccination). Here, ''N''=participants evaluable for this outcome measure. Data was not collected from participants in Groups 7 and 11 as no participants received booster vaccination due to study termination.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 7 and 11 Combined | Group 8 and 10 Combined
Number analyzed (Participants) | 0 | 92
Percentage of participants
  AEs |  | 17.4
  SAEs |  | 2.2
  MAEs |  | 15.2
  NDCMC |  | 0

24. Primary Outcome: Percentage of Participants With AEs, SAEs, MAEs and NDCMC Throughout Booster Stage: Group 7 and 11 Combined Versus Group 8 and 10 Combined
Description: as for outcome 15
Time Frame: From 1 month after booster vaccination up to 6 months after booster vaccination (maximum up to 6 months)
Population: Booster vaccination safety population included participants who received booster dose of investigational product, had safety follow-up between Visit 5 and prior to Visit 6 (after booster vaccination). Here, ''N''=participants evaluable for this outcome measure. Data was not collected from participants in Groups 7 and 11 as no participants received booster vaccination due to study termination.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 7 and 11 Combined | Group 8 and 10 Combined
Number analyzed (Participants) | 0 | 92
Percentage of participants
  AEs |  | 40.2
  SAEs |  | 2.2
  MAEs |  | 25.0
  NDCMC |  | 0

25. Secondary Outcome: hSBA Geometric Mean Titers (GMTs) for Each of the MenB Test Strains: 1 Month After Primary Vaccination 2 in Group 3 and 4 Combined Versus Group 5
Description: GMTs were calculated by exponentiating mean logarithm of titers and CIs were calculated by exponentiating confidence limits based on the Student t distribution for the mean logarithm of the titers.
Time Frame: 1 Month after primary Vaccination 2
Population: Post-primary vaccination 2 evaluable immunogenicity population: participants randomized to study group of interest; eligible through Visit(V)4; received vaccine at V1,V3;blood drawn for assay testing at required timeframes at V4; had at least 1 valid, determinate MenA, MenC, MenW, MenY, or MenB assay result at V4;received no prohibited vaccines/treatment,no protocol deviations through V4. Here,''N''= participants evaluable for the outcome measure;''n''= participants evaluable for specific rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Group 3 and 4 Combined: Group3:Infant participants aged 2 months were administered single IM injection of 0.25mL bivalent rLP2086(60μg) into left thigh,0.5mL Nimenrix into right thigh at Day 1(primary vacc 1),Month 2(primary vacc 2).PLP or SLP administered orally. Participants received single IM injection of 0.25mL bivalent rLP2086(60 μg) into left thigh and 0.5mL Nimenrix into right thigh approx. 10 months after vacc1(booster vacc).Participants received single IM injection of Prevenar 13,Vaxelis into right thigh at 2 and 4 months of age.Group4: Infant participants aged 2 months were administered single IM injection of 0.25 mL bivalent rLP2086(60 μg) into left thigh,0.5 mL Nimenrix into right thigh at Day 1(primary vacc 1) and Month 2(primary vacc 2).Participants received single IM injection of 0.25mL of bivalent rLP2086(60 μg) into left thigh and 0.5 mL of Nimenrix into right thigh approx.10 months after vacc 1(booster vacc).Participants received single IM injection of Prevenar 13,Vaxelis into right thigh at 2 and 4 months of age.
Arm/Group | Group 3 and 4 Combined | Group 5 (120 mcg rLP2086 +Nimenrix +PLP)
Number analyzed (Participants) | 35 | 45
Titers
  PMB80 (A22): number analyzed (Participants) | 30 | 44
  PMB80 (A22) | 13.9 [10.8 to 18.0] | 15.3 [12.1 to 19.3]
  PMB2707 (B44) | 25.0 [19.9 to 31.4] | 25.0 [19.9 to 31.4]

26. Secondary Outcome: hSBA GMTs for Each of the MenB Test Strains: 1 Month After Booster Vaccination in Groups 3, 4 and 5
Description: GMTs were calculated by exponentiating the mean logarithm of the titers and CIs were calculated by exponentiating the confidence limits based on the Student t distribution for the mean logarithm of the titers. No serum samples were collected after booster dose for groups 4 and 5 due to study termination.
Time Frame: 1 month after booster vaccination
Population: Post-primary vaccination 2 evaluable immunogenicity population:eligible participants randomized through Visit(V)4;received vaccine at V1,V3;blood drawn for assay testing within required timeframes at V4;had at least 1 valid, determinate MenA, C, W, Y, or B assay result at V4;received no prohibited vaccines/treatment;no protocol deviation through V4. Here,''N''=participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 3 (60 mcg rLP2086 +Nimenrix +PLP/SLP) | Group 4 (60 mcg rLP2086 +Nimenrix) | Group 5 (120 mcg rLP2086 +Nimenrix +PLP)
Number analyzed (Participants) | 18 | 0 | 0
Titers
  PMB80 (A22) | 21.8 (11.1) [11.1 to 42.6] |  |
  PMB2707 (B44) | 25.4 (12.6) [12.6 to 51.1] |  |

27. Secondary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Each Primary Vaccination: Group 3, 4 and 5
Description: Local reactions included pain at injection site, redness and swelling and were recorded by participant's in an electronic diary (e-diary). Redness and swelling were measured and recorded in caliper units. 1 caliper unit =0.5 centimeter (cm) and graded as mild: >2.0 to 5.0 cm, moderate: >5.0 to 10.0 cm and severe: >10.0 cm. Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfered with daily activity and severe: prevented daily activity. Percentage of participants with local reactions at injection site on left arm were reported in this outcome measure.
Time Frame: Within 7 Days after primary Vaccination(Vac) 1 and 2
Population: Safety population included all randomized participants who received at least 1 dose of investigational product and had safety data reported after vaccination. Here, ''N''=participants evaluable for this outcome measure; ''n''= participants evaluable for specific rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 3 (60 mcg rLP2086 +Nimenrix +PLP/SLP) | Group 4 (60 mcg rLP2086 +Nimenrix) | Group 5 (120 mcg rLP2086 +Nimenrix +PLP)
Number analyzed (Participants) | 36 | 16 | 53
Percentage of participants
  Vaccination 1:Redness:Mild | 27.8 [14.2 to 45.2] | 18.8 [4.0 to 45.6] | 13.2 [5.5 to 25.3]
  Vacc1Redness:Moderate | 8.3 [1.8 to 22.5] | 0 [0.0 to 20.6] | 3.8 [0.5 to 13.0]
  Vacc1Redness: Severe | 0 [0.0 to 9.7] | 0 [0.0 to 20.6] | 0 [0.0 to 6.7]
  Vacc1:Swelling: Mild | 16.7 [6.4 to 32.8] | 6.3 [0.2 to 30.2] | 9.4 [3.1 to 20.7]
  Vacc1:Swelling: Moderate | 11.1 [3.1 to 26.1] | 12.5 [1.6 to 38.3] | 5.7 [1.2 to 15.7]
  Vacc1:Swelling: Severe | 0 [0. to 9.7] | 0 [0.0 to 20.6] | 0 [0.0 to 6.7]
  Vac1Tenderness at inj.site:Mild | 19.4 [8.2 to 36.0] | 12.5 [1.6 to 38.3] | 22.6 [12.3 to 36.2]
  Vac1Tenderness at inj.site: Moderate | 41.7 [25.5 to 59.2] | 18.8 [4.0 to 45.6] | 20.8 [10.8 to 34.1]
  Vac1Tenderness at inj.site: Severe | 0 [0.0 to 9.7] | 0 [0.0 to 20.6] | 1.9 [0.0 to 10.1]
  Vac2Redness: Mild: number analyzed (Participants) | 21 | 16 | 52
  Vac2Redness: Mild | 33.3 [14.6 to 57.0] | 18.8 [4.0 to 45.6] | 19.2 [9.6 to 32.5]
  Vac2Redness: Moderate: number analyzed (Participants) | 21 | 16 | 52
  Vac2Redness: Moderate | 4.8 [0.1 to 23.8] | 0 [0.0 to 20.6] | 3.8 [0.5 to 13.2]
  Vac2Redness: Severe: number analyzed (Participants) | 21 | 16 | 52
  Vac2Redness: Severe | 0 [0.0 to 16.1] | 0 [0.0 to 20.6] | 0 [0.0 to 6.8]
  Vac2Swelling: Mild: number analyzed (Participants) | 21 | 16 | 52
  Vac2Swelling: Mild | 19.0 [5.4 to 41.9] | 12.5 [1.6 to 38.3] | 9.6 [3.2 to 21.0]
  Vac2Swelling: Moderate: number analyzed (Participants) | 21 | 16 | 52
  Vac2Swelling: Moderate | 0 [0.0 to 16.1] | 12.5 [1.6 to 38.3] | 1.9 [0.0 to 10.3]
  Vac2Swelling Severe: number analyzed (Participants) | 21 | 16 | 52
  Vac2Swelling Severe | 0 [0.0 to 16.1] | 0 [0.0 to 20.6] | 0 [0.0 to 6.8]
  Vac2Tenderness at inj.site Mild: number analyzed (Participants) | 21 | 16 | 52
  Vac2Tenderness at inj.site Mild | 28.6 [11.3 to 52.2] | 12.5 [1.6 to 38.3] | 32.7 [20.3 to 47.1]
  Vac2Tenderness at inj.siteModerate: number analyzed (Participants) | 21 | 16 | 52
  Vac2Tenderness at inj.siteModerate | 9.5 [1.2 to 30.4] | 18.8 [4.0 to 45.6] | 17.3 [8.2 to 30.3]
  Vac2Tenderness at inj.siteSevere: number analyzed (Participants) | 21 | 16 | 52
  Vac2Tenderness at inj.siteSevere | 0 [0.0 to 16.1] | 6.3 [0.2 to 30.2] | 1.9 [0.0 to 10.3]

28. Secondary Outcome: Percentage of Participants With Systemic Events and Antipyretic Use Within 7 Days After Each Primary Vaccination: Group 3,4 and 5
Description: Systemic events were recorded by participant's parents/legal guardians in e-diary. Fever was defined as temperature >=38.0 degrees (deg) Celsius(C) and was categorized as 38.0 to 38.4 deg C, >38.4 to 38.9 deg C, >38.9 to 40.0 deg C and >40.0 deg C. Exact 2-sided CI was based on the Clopper and Pearson method. Decreased appetite was categorized as Grade 1:decreased interest in eating, Grade 2:decreased oral intake, Grade3: refusal to feed. Drowsiness: Grade 1 Increased or prolonged sleeping bouts,Grade2: Slightly subdued interfering with daily activity, Grade3; Disabling, not interested in usual daily activity. Irritability; Grade1: Easily consolable, Grade2: requiring increased attention, Grade 3: Inconsolable; crying could not be comforted.
Time Frame: Within 7 Days after primary Vaccination 1 and 2
Population: Primary vaccination 1 safety population included all randomized participants who received the first dose of investigational product at Visit 1 and had safety follow-up between Visit 1 and prior to Visit 3. Here, ''N''=participants evaluable for this outcome measure; ''n''= participants evaluable for specific rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 3 (60 mcg rLP2086 +Nimenrix +PLP/SLP) | Group 4 (60 mcg rLP2086 +Nimenrix) | Group 5 (120 mcg rLP2086 +Nimenrix +PLP)
Number analyzed (Participants) | 36 | 16 | 53
Percentage of participants
  Vac1Fever38.0°C to 38.4°C | 30.6 [16.3 to 48.1] | 18.8 [4.0 to 45.6] | 35.8 [23.1 to 50.2]
  Vac1Fever>38.4°C to 38.9°C | 27.8 [14.2 to 45.2] | 6.3 [0.2 to 30.2] | 17.0 [8.1 to 29.8]
  Vac1Fever>38.9°C to 40.0°C | 0 [0.0 to 9.7] | 0 [0.0 to 20.6] | 11.3 [4.3 to 23.0]
  Vac1Fever >40.0°C | 0 [0.0 to 9.7] | 0 [0.0 to 20.6] | 0 [0.0 to 6.7]
  Vac1Decreased appetite Mild | 25.0 [12.1 to 42.2] | 6.3 [0.2 to 30.2] | 28.3 [16.8 to 42.3]
  Vac1Decreased appetite Moderate | 22.2 [10.1 to 39.2] | 43.8 [19.8 to 70.1] | 34.0 [21.5 to 48.3]
  Vac1Decreasedappetite Severe | 2.8 [0.1 to 14.5] | 0 [0.0 to 20.6] | 3.8 [0.5 to 13.0]
  Vac1IrritabilityMild | 16.7 [6.4 to 32.8] | 6.3 [0.2 to 30.2] | 5.7 [1.2 to 15.7]
  Vac1IrritabilityModerate | 58.3 [40.8 to 74.5] | 75.0 [47.6 to 92.7] | 58.5 [44.1 to 71.9]
  Vac1IrritabilitySevere | 8.3 [1.8 to 22.5] | 6.3 [0.22 to 30.2] | 13.2 [5.5 to 25.3]
  Vac1DrowsinessMild | 36.1 [20.8 to 53.8] | 37.5 [15.2 to 64.6] | 49.1 [35.1 to 63.2]
  Vac1DrowsinessModerate | 33.3 [18.6 to 51.0] | 31.3 [11.0 to 58.7] | 39.6 [26.5 to 54.0]
  Vac1DrowsinessSevere | 2.8 [0.1 to 14.5] | 0 [0.0 to 20.6] | 3.8 [0.5 to 13.0]
  Use of antipyretic medication | 58.3 [40.8 to 74.5] | 56.3 [29.9 to 80.2] | 83.0 [70.2 to 91.9]
  Vac2 >38.0°C to 38.4°C: number analyzed (Participants) | 21 | 16 | 52
  Vac2 >38.0°C to 38.4°C | 23.8 [8.2 to 47.2] | 25.0 [7.3 to 52.4] | 28.8 [17.1 to 43.1]
  Vac2 >>38.4°C to 38.9°C: number analyzed (Participants) | 21 | 16 | 52
  Vac2 >>38.4°C to 38.9°C | 23.8 [8.2 to 47.2] | 25.0 [7.3 to 52.4] | 25.0 [14.0 to 38.9]
  Vac2>>38.9°C to 40.0°C: number analyzed (Participants) | 21 | 16 | 52
  Vac2>>38.9°C to 40.0°C | 4.8 [0.1 to 23.8] | 0 [0.0 to 20.6] | 13.5 [5.6 to 25.8]
  Vac2>40.0°C: number analyzed (Participants) | 21 | 16 | 52
  Vac2>40.0°C | 0 [0.0 to 16.1] | 0 [0.0 to 20.6] | 0 [0.0 to 6.8]
  Vac2Decreased appetiteMild: number analyzed (Participants) | 21 | 16 | 52
  Vac2Decreased appetiteMild | 4.8 [0.1 to 23.8] | 6.3 [0.2 to 30.2] | 28.8 [17.1 to 43.1]
  Vac2Decreased appetiteModerate: number analyzed (Participants) | 21 | 16 | 52
  Vac2Decreased appetiteModerate | 28.6 [11.3 to 52.2] | 50.0 [24.7 to 75.3] | 38.5 [25.3 to 53.0]
  Vac2Decreased appetite Severe: number analyzed (Participants) | 21 | 16 | 52
  Vac2Decreased appetite Severe | 4.8 [0.1 to 23.8] | 6.3 [0.2 to 30.2] | 5.8 [1.2 to 15.9]
  Vac2 Irritability Mild: number analyzed (Participants) | 21 | 16 | 52
  Vac2 Irritability Mild | 28.6 [11.3 to 52.2] | 12.5 [1.6 to 38.3] | 21.2 [11.1 to 34.7]
  Vac2IrritabilityModerate: number analyzed (Participants) | 21 | 16 | 52
  Vac2IrritabilityModerate | 23.8 [8.2 to 47.2] | 68.8 [41.3 to 89.0] | 48.1 [34.0 to 62.4]
  Vac2IrritabilitySevere: number analyzed (Participants) | 21 | 16 | 52
  Vac2IrritabilitySevere | 4.8 [0.1 to 23.8] | 0 [0.0 to 20.6] | 9.6 [3.2 to 21.0]
  Vac2DrowsinessMild: number analyzed (Participants) | 21 | 16 | 52
  Vac2DrowsinessMild | 47.6 [25.7 to 70.2] | 43.8 [19.8 to 70.1] | 40.4 [27.0 to 54.9]
  Vac2DrowsinessModertae: number analyzed (Participants) | 21 | 16 | 52
  Vac2DrowsinessModertae | 23.8 [8.2 to 47.2] | 12.5 [1.6 to 38.3] | 28.8 [17.1 to 43.1]
  Vac2DrowsinessSevere: number analyzed (Participants) | 21 | 16 | 52
  Vac2DrowsinessSevere | 0 [0.0 to 16.1] | 0 [0.0 to 20.6] | 3.8 [0.5 to 13.2]
  Vac2Use of antipyretic medication: number analyzed (Participants) | 21 | 16 | 52
  Vac2Use of antipyretic medication | 81.0 [58.1 to 94.6] | 87.5 [61.7 to 98.4] | 86.5 [74.2 to 94.4]

29. Secondary Outcome: Percentage of Participants With AEs, SAEs, MAEs and NDCMC: Groups 3, 4 and 5
Description: as for outcome 16
Time Frame: Within 30 days after any vaccination
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Group 3 (60 mcg rLP2086 +Nimenrix +PLP/SLP) | Group 4 (60 mcg rLP2086 +Nimenrix) | Group 5 (120 mcg rLP2086 +Nimenrix +PLP)
Number analyzed (Participants) | 36 | 16 | 53
Percentage of participants
  AEs | 52.8 | 68.8 | 60.4
  SAEs | 2.8 | 6.3 | 20.8
  MAEs | 47.2 | 62.5 | 47.2
  NDCMC | 0 | 6.3 | 0

ADVERSE EVENTS:
Time Frame: Systematic assessment(SA): local reactions/systemic events within 7 days after vaccination 1, 2 and booster vaccination; Non-systematic assessment: SAEs and other AEs from Day 1 up to 196 days after last study vaccination (up to 12 months for Group1 and 2; up to 16 months for Group 3,4,5,7,8,10,11)
Description: Same event may appear as both non-SAE and SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE.
Arm/Group | Group 1 (MenABCWY +PLP) | Group 2 (MenABCWY) | Group 3 (60 mcg rLP2086 +Nimenrix +PLP/SLP) | Group 4 (60 mcg rLP2086 +Nimenrix) | Group 5 (120 mcg rLP2086 +Nimenrix +PLP) | Group 7 (MenABCWY +SLP) | Group 8 (Bexsero +Nimenrix +PLP) | Group 10 (Bexsero +Nimenrix) | Group 11 (MenABCWY +TLP)
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/25 | 0/36 | 0/16 | 0/53 | 1/50 | 0/55 | 0/55 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/23 | 1/25 | 1/36 | 1/16 | 11/53 | 5/50 | 1/55 | 6/55 | 1/12
Other Adverse Events (participants affected / at risk) | 23/23 | 25/25 | 36/36 | 16/16 | 53/53 | 50/50 | 54/55 | 55/55 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (MenABCWY +PLP) (N=23) | Group 2 (MenABCWY) (N=25) | Group 3 (60 mcg rLP2086 +Nimenrix +PLP/SLP) (N=36) | Group 4 (60 mcg rLP2086 +Nimenrix) (N=16) | Group 5 (120 mcg rLP2086 +Nimenrix +PLP) (N=53) | Group 7 (MenABCWY +SLP) (N=50) | Group 8 (Bexsero +Nimenrix +PLP) (N=55) | Group 10 (Bexsero +Nimenrix) (N=55) | Group 11 (MenABCWY +TLP) (N=12)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Papilloedema (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sudden infant death syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis bacillus (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Human herpesvirus 7 infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Meningitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (MenABCWY +PLP) (N=23) | Group 2 (MenABCWY) (N=25) | Group 3 (60 mcg rLP2086 +Nimenrix +PLP/SLP) (N=36) | Group 4 (60 mcg rLP2086 +Nimenrix) (N=16) | Group 5 (120 mcg rLP2086 +Nimenrix +PLP) (N=53) | Group 7 (MenABCWY +SLP) (N=50) | Group 8 (Bexsero +Nimenrix +PLP) (N=55) | Group 10 (Bexsero +Nimenrix) (N=55) | Group 11 (MenABCWY +TLP) (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Congenital skin disorder (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Odontogenic cyst (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Plagiocephaly (Congenital, familial and genetic disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Precocious puberty (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 3 | 1 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 0
Gingival cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infantile colic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Teething (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1 | 3 | 0 | 0 | 1 | 2 | 1 | 0
Drug withdrawal syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 6 | 2 | 2 | 0 | 4 | 4 | 3 | 5 | 0
Pyrexia (FEVER) (General disorders) | 15 | 19 | 25 | 10 | 42 | 38 | 32 | 39 | 7
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Swelling (SWELLING) (General disorders) | 10 | 14 | 13 | 5 | 10 | 26 | 30 | 31 | 2
Tenderness (TENDERNESS) (General disorders) | 20 | 20 | 23 | 8 | 35 | 41 | 41 | 45 | 8
Vaccination site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Food allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Milk allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 2 | 4 | 3 | 2 | 2 | 3 | 1 | 3 | 1
Bronchitis (Infections and infestations) | 2 | 2 | 1 | 0 | 1 | 0 | 1 | 1 | 0
Bronchitis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 2 | 3 | 0 | 1 | 4 | 8 | 5 | 6 | 1
Candida nappy rash (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 4 | 3 | 0 | 3 | 3 | 1 | 4 | 4 | 1
Ear infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 6 | 8 | 2 | 0 | 1 | 1 | 4 | 4 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 7 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Herpangina (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Impetigo (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 3 | 2 | 0 | 3 | 2 | 1 | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Mumps (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 5 | 2 | 0 | 1 | 1 | 3 | 3 | 5 | 0
Oral candidiasis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 1 | 4 | 1 | 2 | 0 | 0 | 0 | 2 | 1
Otitis media acute (Infections and infestations) | 4 | 6 | 2 | 1 | 2 | 1 | 1 | 2 | 0
Parvovirus B19 infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 3 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 3 | 0 | 1 | 0 | 0 | 3 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 4 | 5 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Skin candida (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Superinfection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 5 | 6 | 2 | 7 | 7 | 11 | 11 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Vaccination site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 4 | 2 | 0 | 0 | 1 | 0 | 1 | 4 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 3 | 0 | 1 | 1 | 0 | 2 | 3 | 1
Vulvovaginitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 2
Decreased appetite (DECREASED APPETITE) (Metabolism and nutrition disorders) | 18 | 17 | 25 | 11 | 46 | 38 | 37 | 41 | 9
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight gain poor (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acquired plagiocephaly (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
External hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypersomnia (INCREASED SLEEP) (Nervous system disorders) | 18 | 18 | 32 | 12 | 50 | 39 | 44 | 43 | 10
Motor developmental delay (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Irritability (Psychiatric disorders) | 2 | 0 | 0 | 0 | 1 | 4 | 3 | 1 | 2
Irritability (IRRITABILITY) (Psychiatric disorders) | 22 | 20 | 32 | 14 | 50 | 49 | 44 | 49 | 12
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 1 | 1 | 1 | 2 | 2 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema (REDNESS) (Skin and subcutaneous tissue disorders) | 8 | 13 | 18 | 6 | 19 | 22 | 31 | 35 | 4
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 3 | 1 | 0
Viral rash (Infections and infestations) | 0 | 3 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Study was terminated based on Sponsor's careful review of available safety data in concert with the recommendation of an independent Data Monitoring Committee.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT04645966/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/66/NCT04645966/SAP_001.pdf